CLINICAL TRIAL: NCT05931146
Title: Effectiveness of Smartphone Application for Weight Loss in Healthy Female Adults
Brief Title: Effectiveness of Smartphone Application for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REC/01408 Maria Mishal
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Weight Loss
Keywords: Adult Females; Exercise Adherence; Obesity; Physical Activity; VO2 Max; Weight Loss
MeSH Terms: conditions — Weight Loss; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MyNetDiary app group (Experimental): Smart phone application MyNetDiary will be used to track calories and exercise log. The intervention period would last for 3 months.
  Interventions: Other: MyNetDiary app group
- Paper diary group (Experimental): This group will follow paper diary to track calories and exercise log for 3 months.
  Interventions: Other: Paper diary group

INTERVENTIONS:
Other: MyNetDiary app group — MyNetDiary will be used to track calories, and exercise while motivating for living a healthier life each day.The intervention period would last for three months. Total energy expenditure (TEE) of every participant enrolled into the study would be calculated at the start of the study and an exercise and diet plan with a calorie deficit of around 1000 kcal per week would be provided to the participant. The diet and exercise plan would be modified according to the new TEE of the participant. MyNetDiary app has built-in food and exercise activities with their respective calories' count. Moreover, customized foods and exercises can also be added into the application
  Arms: MyNetDiary app group
Other: Paper diary group — Paper Diary will be used to track calories and exercise. The nutritional intake and exercise would be recorded for three months. The diet and exercise plans would be modified according to the new Total Energy Expenditure of the participants.
  Arms: Paper diary group

SUMMARY:
The aim of this study is

To determine the effectiveness of smartphone application for weight loss in healthy female adults.

To determine the association between fitness application usage and physical activity behavior of the healthy female adults.

DETAILED DESCRIPTION:
Obesity has turned into a significant, rising well-being epidemic around the world. Doing almost no physical work has been connected with chronic weakness results and diminished personal satisfaction in adulthood. It has been perceived that innovation can uphold wellbeing upgrades around the world. The applications that target wellbeing advancement have turned into a focal piece of individuals' lives and have exhibited enormous expansions being used. Proper evidence behind usage of smart phone application for weight loss is sparse and is based on different clinical experiences and a smaller number of studies with limited methodological design. This study will contribute to describing the effectiveness of smartphone application for weight loss in female adults as well as to determine the association between fitness application usage and physical activity behavior.

ELIGIBILITY:
Inclusion Criteria:

* Adult females
* Age between 18-40 years.
* Individuals with BMI ≥ 25

Exclusion Criteria:

* Pathological conditions affecting any system
* Suffering from recent unhealed MSK injury/Trauma

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Weight | 3 months
  It is the estimation of weight without wearing extra things by the individual. Excess or reduced weight is viewed as a sign of deciding an individual's health, with body volume estimation giving an additional aspect by calculating the distribution of body weight. A weight machine is usually used for this purpose. Weight machine is a gadget used to measure weight or mass, which is also called weight scale and weight balance system. The conventional scale comprises of two plates suspended at equal distances from a fulcrum. However, in this study, a digital weight machine will be used. The hardware comprises of a load cell or a weighing scale. The load cell calculates the person's weight and turns the mechanical force into electrical signals that can be easily obtained after microcontroller processing. Excess or reduced weight is viewed as a sign of deciding an individual's health, with body volume estimation giving an additional aspect by calculating the distribution of body
BMI | 3 months
  BMI stands for Body Mass Index. Mathematically it is calculated as, an individual's weight in kilograms (or pounds) divided by the square of level in meters (or feet). The categories of BMI are as follows: < 18.5 as underweight, 18.5 < 25 as normal weight, BMI 25 < 30 as overweight, BMI 30 < 35 as low obesity, BMI 35 < 40 as medium obesity and BMI ≥ 40 as extreme obesity

SECONDARY OUTCOMES:
MyNetDairy App | 3 months
  The app usage data will be collected from the phone with the help of phone's app usage record and daily usage of app, its exercise log and diet log would be recorded to maintain app usage data.
Level of physical activity | 3 months
  The physical activity level is a method for communicating an individual's day to day activity as a number and is utilized to gauge an individual's energy consumption
Exercise adherence | 3 months
  Exercise adherence is a term used to define how well a patient or client is following their home exercise program or gym program and the suggestions made to them by their health expert or fitness coach. This would be recorded with the help of daily exercise and diet log by using diary or app usage.
Blood Pressure | 3 months
  Blood pressure is the force of blood pushing against the walls of arteries. Each time heart beats, it siphons blood into the supply routes. Blood pressure is highest when heart beats, pumping the blood. This is called systolic pressure. At the point when heart is very still, between beats, blood pressure falls. This is called diastolic pressure. Sphygmomanometer is used to measure blood pressure. It typically consists of an inflatable rubber cuff which is applied to the arm and connected to a column of mercury next to a graduated scale, enabling the determination of systolic and diastolic blood pressure by increasing and gradually releasing the pressure in the cuff. Normal blood pressure is considered as 120/80 mmHg as systolic/diastolic pressure.
VO2 max | 3 months
  It is the highest rate of oxygen consumption attainable during maximal exercise

CONTACTS AND LOCATIONS:
Overall Officials: Noman Sadiq, MS-SPT, Principal Investigator — Riphah International University, Islamabad.
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No